CLINICAL TRIAL: NCT06186960
Title: Tandem VR: Synchronized Nature-Based Experiences in Virtual Reality for Hospice Patients and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2079177-3
Record Dates: First submitted 2023-11-30; First posted 2024-01-02 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-01

CONDITIONS: Hospice; End of Life; Palliative Care; Pain; Anxiety; Fear of Death
Keywords: hospice; palliative care; virtual reality; VR; quality of life; personalized; nature; tandem
MeSH Terms: conditions — Death; Pain; Anxiety Disorders; Necrophobia

STUDY DESIGN:
Intervention Model Description: Multiple Method Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tandem Virtual Reality Experience (Experimental): Tandem VR Intervention After the surveys are completed, the researchers will share a personalized library of immersive, nature-based, 360-degree VR experiences for the participant-caregiver dyads to choose from based on their VR Intake Form. Once the dyad has determined their desired Tandem VR experience from the library, the researchers will assist the dyads in donning the VR head mounted display (HMD). The researchers will ensure the safety of both dyads while using the HMDs. The researchers will then initiate the Tandem VR experience. The duration of the Tandem VR experience will be 5-15 minutes.
  Interventions: Device: Tandem Virtual Reality

INTERVENTIONS:
Device: Tandem Virtual Reality — Hospice patients and their primary caregiver will each wear virtual reality headsets and will experience a customized and synchronized 5-15min virtual reality experience.

SUMMARY:
Background: Nature-based virtual reality (VR) and other outdoor experiences in head-mounted displays (HMDs) offer powerful, non-pharmacological tools for hospice teams to help patients undergoing end-of-life (EOL) transitions. However, the psychological distress of the patient-caregiver dyad is interconnected and highlights the interdependence and responsiveness to distress as a unit. Hospice care services and healthcare need strategies to help patients and informal caregivers with EOL transitions.

DETAILED DESCRIPTION:
Methods: This study uses a synchronized Tandem VR approach where patient- caregiver dyads experience immersive nature-based and other outdoor VR content. This mixed methods study will recruit 20 patient-caregiver dyads (N = 40) enrolled in home hospice services nearing the end-of-life. Dyads will experience a personalized nature-based or other outdoor VR experience lasting 5-15 minutes. Self-reported questionnaires and semi-structured interviews will be collected before and after the VR intervention to identify the impacts of personalized nature-based and other outdoor Tandem VR experiences on the QOL, pain, and fear of death in patient-caregiver dyads enrolled with hospice services. Additionally, this protocol will determine the acceptance of personalized nature-based and other outdoor Tandem VR experiences by dyads as a non-pharmacological modality for addressing patient and caregiver needs. Acceptance was quantified by the number of dyads accepting or declining the VR experience during recruitment.

Discussion: Using personalized, nature-based and other outdoor VR experiences, the patient-caregiver dyads can simultaneously engage in an immersive encounter to help alleviate symptoms associated with declining health and EOL phases for the patient and the often overburdened caregiver. This protocol focuses on meeting the need for person- and caregiver-centered, non-pharmacological interventions to reduce physical, psychological, and spiritual distress.

ELIGIBILITY:
Inclusion criteria:

* English speaking
* Projected life expectancy of <6 months (established by hospice experts)
* Cognitively intact (has sufficient judgment, planning, organization, and self-control)

Exclusion criteria:

* Having a cognitive impairment that affects protocol participation. This will be done with the assistance of Research Recruiters to assess eligibility.
* Have a condition that interferes with VR usage, including but not limited to seizures, facial injury precluding safe placement of headset
* Have a prognosis of hours or actively dying at the time enrollment
* Patients with motion sickness
* Patients with claustrophobia
* Patients with visual and hearing impairment
* Patients with inability to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Quality of life (QOL) | Up to 12 months
  Quality of life will be measured with the McGill Quality of Life Questionnaire (MQOL-E). This assesses eight important life domains: cognition, healthcare, environment, feeling like a burden, and their relationships with physical, psychological, social, and existential/spiritual domains. The 16-item questionnaire uses a 0-10 response scale with a higher score indicating a higher quality of life.
Fear of Death | Up to 12 months
  The Collett-Lester Fear of Death Scale (CL-FODS), measures changes in perception of fear of death and 28 items. The CL-FODS uses a 5-Likert scale ranging from 1= not to 5=very for how disturbed or made anxious a person is by different aspects of death and dying. A higher score indicates a higher fear of death. Some example items include rating how disturbed or made anxious you are about the shortness of life, the lack of control over dying, and feeling lonely without your person. The CL-FODS has four subsections: Death of Self, Death of Others, Dying of Self, and Dying of Others. The means of each subsection and then the total scale scores illustrate the degree of anxiety about death and dying, with a higher value indicating the severity of anxiety about death and dying.
Perception of Pain | Up to 12 months
  Wisconsin Brief Pain Scale Questionnaire will assess perception of pain. Patients will rate their pain from 0=no pain to 10=worst pain imaginable in response to items such as "average pain," "worst pain," "least pain" over the last seven days, and "pain right now." An average of the responses to these items is used to create a single pain severity score. A higher score indicates more perceptions of pain.
Acceptance of Tandem VR | Up to 12 months
  Determine the acceptance of personalized nature-based Tandem VR experiences by dyads as a non-pharmacological modality for addressing the needs of dyads. Acceptance is quantified by the number of dyads accepting or declining the VR experience during recruitment.
Perceived benefits and value of Tandem VR | Up to 12 months
  Semi-structured interview data will be gathered and examined using a thematic analysis to capture the perceived benefits and value of Tandem VR.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua K Pope, Principal Investigator — Prisma Health Hospice of the Foothills
Locations (1):
- Cottingham Hospice House, Seneca, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McAnirlin O, Thrift J, Li F, Pope JK, Browning MHEM, Moutogiannis PP, Thomas G, Farrell E, Evatt MM, Fasolino T. The Tandem VR protocol: Synchronized nature-based and other outdoor experiences in virtual reality for hospice patients and their caregivers. Contemp Clin Trials Commun. 2024 Jun 22;40:101318. doi: 10.1016/j.conctc.2024.101318. eCollection 2024 Aug. PMID 39045392

DOCUMENTS (1):
  • Informed Consent Form (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT06186960/ICF_000.pdf